CLINICAL TRIAL: NCT01786031
Title: Prostate Cancer Evaluation of TaRgets in Genito Urinary Screening Program
Acronym: PETRUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00668-35
Record Dates: First submitted 2012-12-03; First posted 2013-02-07 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Castration Resistant Prostate Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): metastasis biopsy
  Interventions: Other: metastasis biopsy

INTERVENTIONS:
Other: metastasis biopsy

SUMMARY:
Toward personalised treatment in early metastatic prostate cancer based on the assessment of biomarkers in cancer tissue samples and circulating tumour cells.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer patients
* Castration Resistant
* Prostatic tissue available
* Metastasis which may be biopsied

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Biomarker | assessed at the end of recruitment, up to 2 years
  success to evaluate at least one molecular analysis in tumor tissues (prostate and/or metastatic site) AND in CTC

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Lindsay CR, Le Moulec S, Billiot F, Loriot Y, Ngo-Camus M, Vielh P, Fizazi K, Massard C, Farace F. Vimentin and Ki67 expression in circulating tumour cells derived from castrate-resistant prostate cancer. BMC Cancer. 2016 Feb 29;16:168. doi: 10.1186/s12885-016-2192-6. PMID 26923772